CLINICAL TRIAL: NCT03984487
Title: Pilot RCT of a Daily Living Skills Intervention for Adolescents With Autism Spectrum Disorder in the Last 2 Years of High School
Brief Title: Daily Living Skills Intervention for Adolescents With Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CIN-DUNCAN-2018-2886
Record Dates: First submitted 2019-05-24; First posted 2019-06-13 (Actual); Results first posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial - A study in which the participants are divided by chance into separate groups that compare different treatments or other interventions.
Who Masked: Outcomes Assessor
Masking Description: Coordinator who is assessing goals of participants id masked from knowing which group each participant was randomized to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STRW (Experimental): Participants will receive the daily living skills intervention, Surviving and Thriving in the Real World (STRW).
  Interventions: Behavioral: Surviving and Thriving in the Real World
- PEERS (Active Comparator): Participants will receive a social skills intervention, Program for the Education and Enrichment of Relational Skills (PEERS).
  Interventions: Behavioral: Program for the Education and Enrichment of Relational Skills

INTERVENTIONS:
Behavioral: Surviving and Thriving in the Real World — The STRW intervention consists of 14 weekly concurrent adolescent and parent group sessions. The DLS to be targeted in the intervention include: Morning Routine (i.e., completing a morning personal hygiene routine); Laundry (i.e., sorting clothing, using a washing machine and dryer, and folding and putting clothes away); Kitchen/Cooking (i.e., cooking items in the microwave, oven, and stove, safe kitchen practices, cleaning up the kitchen after cooking, and grocery shopping); Self-Management (i.e., managing worry and stress related to learning DLS and transitioning to adulthood); and Money Management (i.e., using money to purchase items, evaluating the quality and price of items, understanding and using a checking and savings account, and budgeting money to cover expenses).
  Arms: STRW
Behavioral: Program for the Education and Enrichment of Relational Skills — PEERS is an evidence-based social skills training program for youth with social challenges between the ages of 13-18.The program includes a teen group and a parent group that meet concurrently. Teens learn about conversations, electronic communication, joining groups, humor, handling teasing and disagreements, and planning get-togethers with other teens. Parents learn how to coach their teens to continue to use the skills when the program is complete.
  Arms: PEERS

SUMMARY:
The main objective of the current proposal is to conduct a pilot RCT (i.e., treatment group and social skills control group) to examine how participation in Surviving and Thriving in the Real World (STRW) Intervention affects proximal outcomes with a larger sample size (n = 72). As social skills, executive functioning, and parenting factors have been linked to the acquisition of Daily Living Skills (DLS), the current study will also explore how these are linked to participation in STRW. Lastly, goal attainment scaling (GAS) will be utilized, along with gold standard parent report and adolescent self-report measures, to assess DLS.

DETAILED DESCRIPTION:
Individuals with high functioning autism spectrum disorder (ASD) are not developing the skills necessary to successfully transition from adolescence to college, employment, and independent living.

Daily living skills have been linked to positive adult outcome in individuals with ASD.

Despite the importance of daily living skills to adult outcome, adolescents with high functioning ASD have impaired daily living skills.

A complex set of environmental, individual, and family factors likely affect the ability of adolescents with high functioning ASD to acquire critical daily living skills.

There are currently no evidence-based daily living skills intervention packages for adolescents with high functioning ASD that would prepare them for independence in adulthood.

The pilot RCT will consist of running 4 cohorts of 16-20 high functioning adolescents with ASD (IQ>70) and their parents in a STRW treatment group or social skills control group. Once an eligible cohort of 16-20 adolescents with ASD has been recruited, adolescents will be randomly assigned to either the STRW group or control group using a stratified randomized block design with IQ as a strata variable (IQ<85 and IQ>85) to ensure balanced group assignment for each cohort. Approximately 8-10 adolescents with ASD and their parents will participate in each STRW group. Thus, across 4 cohorts, the goal will be to enroll at least a total of 72 adolescents in the study, 36 in the STRW group and 36 in the control group across Years 1-3.

To test Aim 1: Initially a two-sample t-test will be used to test the difference on the change scores in the Vineland-3 DLS domain and GAS (post-treatment and baseline) between the STRW and control groups. Although this is a randomized study it is possible that some of the demographic variables might be differentially distributed between the groups. In this case, the initial analysis will be followed by a general linear regression analysis where cohort will be treated as the main effect and other differentially distributed variables will be added to the model as possible confounders in order to investigate the independent effect of the intervention group on outcome.

To test Aim 2: The within-subject change between post-treatment and 6-month follow-up for each individual receiving the intervention will be calculated and a paired t-test will be conducted to evaluate this change (post-treatment and 6-month follow-up).

To test Aim 3: Exploratory analyses will be conducted to examine the relationship between progress in DLS and executive functioning, social skills, and parenting and family factors. A regression analysis will be used to estimate and examine this potential relationship. In this model the change score (post-treatment and baseline) will be modeled as a function of each of the measures of executive function, social skills and parenting and family factors. This will allow us to characterize the response profile.

ELIGIBILITY:
Inclusion Criteria:

* in the last 2 years of high school
* diagnosis of ASD based on clinical judgement and/or meeting the cut-off score on the Autism Diagnostic Observation Schedule, 2nd Edition
* full scale IQ of 70 or above as measured by the Stanford Binet Intelligence Scales, 5th Edition
* deficient Daily Living Skills as assessed by the Vineland Adaptive Behavior Scales, 3rd Edition - at least 1 of the 3 Daily Living Skills subdomains is at least 15 points below their full scale IQ

Exclusion Criteria:

* significant aggressive behaviors or mental health issues that require treatment out of the scope of the current intervention.
* if the adolescent has already completed the social skills group (PEERS), either at Cincinnati Children's or in another setting, unless it has been a significant amount of time since they did the PEERS group (2-3 years, or up to the discretion of the PI).

Ages: 15 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 73 (Actual)
Dates: Start 2018-05-17 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amie M Duncan, Ph.D., Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited using flyers via our hospital's outpatient autism clinic, research databases, and within the community.
Pre-assignment Details: We had several screen fails, which we compensated for by enrolling above our target number for completion.
  Randomization was stratified based on IQ (i.e., IQ>85 and IQ<85).
Period: Overall Study
Arm/Group | STRW | PEERS
Started | 36 | 37
Completed | 31 | 30
Not Completed | 5 | 7

BASELINE CHARACTERISTICS:
Population: STRW: 36 allocated to intervention, 2 lost to follow up before intervention completion, 3 lost to follow up post-intervention (31 analyzed).
  PEERS: 37 allocated to intervention, 7 lost to follow up before intervention completion (30 analyzed).
Groups:
- Total: Total of all reporting groups
Arm/Group | STRW | PEERS | Total
Number analyzed (Participants) | 36 | 37 | 73
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 36 | 37 | 73
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 11 | 19
  Male | 28 | 26 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 6
  Not Hispanic or Latino | 34 | 32 | 66
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 5 | 10
  White | 28 | 28 | 56
  More than one race | 3 | 2 | 5
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 36 | 37 | 73
IQ [Count of Participants; unit: Participants]
  IQ <70 | 36 | 37 | 73
  IQ >70 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Vineland Adaptive Behavior Scales, 3rd Edition
Description: The VABS-3 is a well-established standardized measure of adaptive behavior that assesses skills in the Communication, Daily Living Skills, and Socialization domains. The Daily Living Skills domain is comprised of the Personal, Domestic, and Community subdomains and has items that directly correspond to goals being targeted in the STRW intervention.
  We are reporting the average (mean) Daily Living Skills Domain Raw Scores, both at baseline at post-treatment. The range for total raw score for the entire domain is 0 to 286.
  The higher the score, the more independent they are at overall daily living skills.
Time Frame: 4 months (from baseline to post-intervention)
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | STRW | PEERS
Number analyzed (Participants) | 31 | 30
Score on a scale
  DLS Domain Raw Scores - Baseline | 195.7 (4.6) | 201.7 (4.7)
  DLS Domain Raw Scores - Post-treatment | 232.2 (4.4) | 227.9 (4.4)

ADVERSE EVENTS:
Time Frame: anywhere from 1 year to 16 months per participant, depending on which intervention they were randomized to (groups were run consecutively, not concurrently).
Description: Definition does not differ from CT. gov.
Arm/Group | STRW | PEERS
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/30
Serious Adverse Events (participants affected / at risk) | 1/31 | 0/30
Other Adverse Events (participants affected / at risk) | 0/31 | 0/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | STRW (N=31) | PEERS (N=30)
Self Injury (Psychiatric disorders) | 1 (1) | 0 (0) — 10/21/2019 - Pt took knife from kitchen drawer during group session and attempted to cut forearm. The wound was superficial and not life-threatening.
Inpatient stay (Psychiatric disorders) | 1 (1) | 0 (0) — Participant was admitted to in-patient psychiatric ward until 12/4/19 for cutting.

LIMITATIONS AND CAVEATS:
Limitations of the current study include use of a caregiver report measure for the primary outcome, a relatively small sample size, and the need for a more diverse sample of autistic teens.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-23): https://cdn.clinicaltrials.gov/large-docs/87/NCT03984487/Prot_SAP_000.pdf
  • Informed Consent Form (2022-12-08): https://cdn.clinicaltrials.gov/large-docs/87/NCT03984487/ICF_001.pdf